CLINICAL TRIAL: NCT03506113
Title: GRam Stain-guided Antibiotics ChoicE for Ventilator-Associated Pneumonia (GRACE-VAP) Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Osaka General Medical Center (Other)
Collaborators: Chukyo Hospital (Unknown); Ebina General Hospital (Unknown); Hitachi General Hospital (Unknown); Kansai Medical University (Other); Kansai Medical University Medical Center (Unknown); Nagasaki University (Other); Saga University (Other); University of the Ryukyus (Other); Wakayama Medical University (Other); Tajima Emergency and Critical Care Medical Center (Unknown); Sapporo City General Hospital (Unknown)
Responsible Party: Principal Investigator, Jumpei Yoshimura, MD, Dr., Osaka General Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29-C0707; UMIN000031933 (Registry Identifier: University hospital Medical Information Network)
Record Dates: First submitted 2018-03-29; First posted 2018-04-23 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Gram staining; Antimicrobial therapy; Empirical therapy; Nosocomial infection; Mechanical ventilation; Intensive care; Sepsis
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Cross Infection; Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gram stain-guided therapy group (Active Comparator): The results of Gram staining of endotracheal aspirate are used to guide the selection of antibiotics. The results of the Gram stains are categorised as Gram-positive cocci (GPC) chains, GPC clusters, Gram-positive bacilli (GPB), Gram-negative rods (GNR), or a combination of these. A non-pseudomonal beta-lactam antibiotic is selected when the Gram stain of the endotracheal aspirate shows only GPC chains and/or GPB. An anti-MRSA agent is selected when the Gram stain results show GPC clusters without GNR. An anti-pseudomonal agent is selected when the Gram stain results show GNR without GPC clusters. The combination of an anti-pseudomonal agent and an anti-MRSA agent is selected when the Gram stain results show both GPC clusters and GNR.
  Interventions: Drug: Gram stain-guided antibiotic choice
- Guidelines-based therapy group (Active Comparator): Patients are administered the combination of an anti-pseudomonal agent and anti-MRSA agent according to the Infectious Disease Society of America and the American Thoracic Society (IDSA/ATS) guidelines because 47.7% of S. aureus isolates are MRSA in Japanese ICUs
  Interventions: Drug: Guidelines-based antibiotics choice

INTERVENTIONS:
Drug: Gram stain-guided antibiotic choice — The results of Gram staining of endotracheal aspirate are used to guide the selection of antibiotics.
  Arms: Gram stain-guided therapy group
Drug: Guidelines-based antibiotics choice — Patients are administered the combination of an anti-pseudomonal agent and anti-MRSA agent according to IDSA/ATS guidelines
  Arms: Guidelines-based therapy group

SUMMARY:
Background: Optimising the use of antibiotic agents is a pressing challenge to overcoming the rapid emergence and spread of multidrug-resistant pathogens in intensive care units (ICUs). Although Gram staining may possibly provide immediate information for predicting pathogenic bacteria, Gram stain-guided initial antibiotic treatment is not well established in the ICU setting. The investigators planned the GRam stain-guided Antibiotics ChoicE for Ventilator-Associated Pneumonia (GRACE-VAP) trial to investigate whether Gram staining can safely restrict the use of broad-spectrum antibiotics in patients with ventilator-associated pneumonia (VAP), which is one of the most common hospital-acquired infections in ICUs.

Methods/Design: The GRACE-VAP trial is a multicenter, randomised, open-label parallel-group trial to assess the non-inferiority of Gram stain-guided initial antibiotic treatment to guidelines-based initial antibiotic treatment for the primary endpoint of clinical cure rate in patients with VAP. Secondary endpoints include the coverage rates of initial antibiotic therapies, the selected rates of anti-pseudomonal agents and anti-methicillin-resistant Staphylococcus aureus (MRSA) agents as initial antibiotic therapies, 28-day all-cause mortality, ICU-free days, ventilator-free days, and adverse events. Participants are randomly assigned to receive Gram stain-guided treatment or guidelines-based treatment at a ratio of 1:1. In the Gram stain group, results of Gram staining of endotracheal aspirate are used to guide the selection of antibiotics. In the guidelines group, the combination of an anti-pseudomonal agent and anti-MRSA agent are administered. A total sample size of 200 was estimated to provide a power of 80% with a 1-sided alpha level of 2.5% and a non-inferiority margin of 20%, considering 10% non-evaluable participants.

Discussion: The GRACE-VAP trial is expected reveal whether Gram staining can reduce the use of broad-spectrum antibiotics without impairing patient outcomes and thereby provide evidence for an antibiotics selection strategy in patients with VAP.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mechanical ventilation in the ICU
* Patients undergoing mechanical ventilation for at least 48 hours
* Patients diagnosed as having VAP, which is defined by a modified clinical pulmonary infection score of 5 or more

Exclusion Criteria:

* Patients having an allergy to study medications
* Pregnant patients
* Patients discharged from ICU
* Patients diagnosed as having heart failure or atelectasis
* Patients administered antibiotics for more than 24 hours when they meet the inclusion criteria
* Patients declined to provide full life support
* Patients judged as inappropriate at the discretion of the study physician.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Clinical cure of VAP | up to 22 days
  Cure is defined as completion of antibiotic therapy within 14 days, improvement or lack of progression of baseline radiographic findings at the end of therapy (EOT), and resolution of signs and symptoms of pneumonia at the follow-up/test of cure visit (FU/TOC) conducted 7 days after EOT. Failure is defined as administration of study medication for 15 days or more, progression of radiological signs of pneumonia at EOT, or relapsed pneumonia at FU/TOC.

SECONDARY OUTCOMES:
Select of anti-pseudomonal agents as initial antibiotic therapies | on day 1
Select of anti-MRSA agents as initial antibiotic therapies | on day 1
Coverage of initial antibiotic therapies | on day 1
  Therapies will be considered appropriate when all pathogens isolated with at least 1+ semi-quantitative growth from endotracheal aspirates are covered by the selected antibiotic agents.
28-day mortality | up to 28 days
ICU-free days | up to 28 days
Ventilator-free days | up to 28 days
Duration of antibiotic therapies | up to 28 days
Need of escalation or de-escalation of antibiotic therapies | up to 28 days
  The investigators evaluate whether antibiotic agents are changed during the treatments of VAP.
Adverse events related to antibiotics | up to 7 days after the end of therapy
  renal impairment, thrombocytopenia, diarrhoea, Clostridium difficile infection, skin rash, and seizure
Inflammation marker | up to 14 days
  Laboratory marker of inflammation (CRP, PCT) on 2, 4, 6, 8, and 14 days
Organ failure control | up to 14 days
  The investigators evaluate Sequential Organ Failure Assessment (SOFA) score on 2, 4, 6, 8, and 14 days. The SOFA score is made of 6 variables, each representing an organ system ( respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems). Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure). The total SOFA score is calculated by the sum of each 6 variables (range, 0-24).
Renal function | up to 14 days
  The investigators evaluate whether participants are performed a renal replacement therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jumpei Yoshimura, MD, Principal Investigator — Osaka General Medical Center; Kazuma Yamakawa, MD, PhD, Study Director — Osaka General Medical Center; Takeshi Morimoto, MD, PhD, MPH, Study Director — Hyogo Medical University
Locations (12):
- Japan (12):
  - Chukyo Hospital, Nagoya, Aichi-ken
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Tajima Emergency and Critical Care Medical Center, Toyooka, Hyōgo
  - Hitachi General Hospital, Hitachi, Ibaraki
  - Ebina General Hospital, Ebina, Kanagawa
  - University of the Ryukyus Hospital, Nishihara, Okinawa
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kansai Medical University Medical Center, Moriguchi, Osaka
  - Nagasaki University Hospital, Nagasaki
  - Osaka General Medical Center, Osaka
  - Saga University Hospital, Saga
  - Wakayama Medical University Hospital, Wakayama

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yoshimura J, Yamakawa K, Ohta Y, Nakamura K, Hashimoto H, Kawada M, Takahashi H, Yamagiwa T, Kodate A, Miyamoto K, Fujimi S, Morimoto T. Effect of Gram Stain-Guided Initial Antibiotic Therapy on Clinical Response in Patients With Ventilator-Associated Pneumonia: The GRACE-VAP Randomized Clinical Trial. JAMA Netw Open. 2022 Apr 1;5(4):e226136. doi: 10.1001/jamanetworkopen.2022.6136. PMID 35394515
- [Derived] Yoshimura J, Yamakawa K, Kinoshita T, Ohta Y, Morimoto T. GRam stain-guided Antibiotics ChoicE for Ventilator-Associated Pneumonia (GRACE-VAP) trial: rationale and study protocol for a randomised controlled trial. Trials. 2018 Nov 8;19(1):614. doi: 10.1186/s13063-018-2971-2. PMID 30409160